## Evaluation of Gingival Crevicular Fluid and Saliva SOST and TWEAK, Gingival Crevicular Fluid RANKL and OPG Levels in Smokers and Non-smokers with Periodontitis

14.09.2023

Statistical analyzes were performed with Jamovi (Version 2.3.24.0) and JASP (Version 0.17.1) programs, and 0.05 (p-value) was taken into account as the significance level in statistical analyses.

While summarizing the study data, "median, minimum and maximum" values were added to the table depending on the distribution for continuous (numerical) variables. Categorical variables were presented as numbers. Normal distribution of numerical variables was evaluated using Shapiro-Wilk, Kolmogorov-Smirnov and Anderson-Darling tests.

To compare categorical variable differences between groups, Pearson Chi-Square test was used in 2x2 tables with expected number of observations being 5 or more, and Fisher's Exact Test was used in tables with expected number of observations below 5. Fisher Freeman Halton test was used in RxC tables with expected number of observations below 5.

When two independent groups were compared, Mann Whitney U test was used in cases where numerical variables were not normally distributed.

When multiple independent groups were compared, the Kruskal-Wallis H test was used when numerical variables were not normally distributed. Differences between groups were evaluated with the Dwass-Steel-Critchlow-Fligner test.

In examining the relationships between numerical variables, Spearman's Rho correlation coefficient was used in cases where the variables were not normally distributed.